CLINICAL TRIAL: NCT04216589
Title: A Single-Arm, Open-Label, Pilot Study of Semaglutide for Non-Alcoholic Fatty Liver Disease (NAFLD), a Metabolic Syndrome With Insulin Resistance, Increased Hepatic Lipids, and Increased Cardiovascular Disease Risk (The SLIM LIVER Study)
Brief Title: Study of Semaglutide for Non-Alcoholic Fatty Liver Disease (NAFLD), a Metabolic Syndrome With Insulin Resistance, Increased Hepatic Lipids, and Increased Cardiovascular Disease Risk (The SLIM LIVER Study)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACTG A5371; 38453 (Registry Identifier: DAIDS-ES Registry Number); NCT05654051 (obsolete NCT alias)
Record Dates: First submitted 2019-12-30; First posted 2020-01-02 (Actual); Results first posted 2024-05-17 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: HIV Infections; Non-Alcoholic Fatty Liver Disease
Keywords: NAFLD; HIV; semaglutide
MeSH Terms: conditions — HIV Infections; Non-alcoholic Fatty Liver Disease | interventions — semaglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Semaglutide (Experimental): All participants received a dose of 0.25 mg of semaglutide weekly starting at study entry, followed by 0.5 mg weekly starting at Week 2, and then 1.0 mg weekly from Weeks 4 through 24.
  Interventions: Drug: Semaglutide

INTERVENTIONS:
Drug: Semaglutide — Administered subcutaneously

SUMMARY:
The purpose of this study was to evaluate the effects of semaglutide on intra-hepatic triglyceride (IHTG) content in people living with HIV (PLWH), central adiposity, insulin resistance or pre-diabetes, and hepatic steatosis.

DETAILED DESCRIPTION:
This study evaluated the effects of semaglutide on intra-hepatic triglyceride (IHTG) content in people living with HIV (PLWH), central adiposity, insulin resistance or pre-diabetes, and hepatic steatosis.

All participants received semaglutide subcutaneously once weekly for 24 weeks, followed by 24 weeks of observation off of the study drug. IHTG was quantified by magnetic resonance imaging-proton density fat fraction (MRI-PDFF) evaluations at two time points during the study.

Participants attended several study visits through Week 48. Participants completed food diaries, adherence and strength assessments, and report on hypoglycemia, vision changes, physical activity, diet, quality of life, and acceptability of study drug. Blood was collected at all visits and stool samples at two visits.

Participants remained on their non-study-provided antiretroviral therapy (ART) throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection, documented by any licensed rapid HIV test or HIV enzyme or chemiluminescence immunoassay (E/CIA) test kit at any time prior to study entry and confirmed by a licensed Western blot or a second antibody test by a method other than the initial rapid HIV and/or E/CIA, or by HIV-1 antigen, plasma HIV-1 RNA viral load.

  * NOTE: The term "licensed" refers to a US Food and Drug Administration (FDA)-approved kit, which is required for all investigational new drug (IND) studies, or for sites located in countries other than the United States, a kit that has been certified or licensed by an oversight body within that country and validated internally. Non-US sites are encouraged to use US FDA-approved methods for IND studies.
  * WHO (World Health Organization) and CDC (Centers for Disease Control and Prevention) guidelines mandate that confirmation of the initial test result must use a test that is different from the one used for the initial assessment. A reactive initial rapid test should be confirmed by either another type of rapid assay or an E/CIA that is based on a different antigen preparation and/or different test principle (e.g., indirect versus competitive), or a Western blot or a plasma HIV-1 RNA viral load.
* Two separate reports of HIV-1 RNA measurements <50 copies/mL, and no HIV-1 RNA measurement >500 copies/mL, during the 48 weeks prior to entry. One of the HIV-1 RNA values must be the screening visit value, and the other value obtained between 24 and 48 weeks prior to entry.

  * NOTE: All values must have been reported from a US laboratory that has a Clinical Laboratory Improvement Amendments (CLIA) certification or its equivalent, or at any network-approved non-US laboratory that is Virology Quality Assurance (VQA) certified.
* No change in antiretroviral therapy (ART) in the 24 weeks prior to entry.

  * NOTE A: Modifications of ART formulation (e.g., from standard formulation to fixed dose combination or single tablet regimen) will be permitted.
  * NOTE B: Within-class substitutions are not permitted.
* No plan to change ART for the study duration.
* Within 30 days prior to pre-entry, a minimum WC measurement of ≥95 cm for individuals assigned male sex at birth or ≥94 cm for individuals assigned female sex at birth.

  * NOTE: For transgender study participants, sites should use the parameter that matches sex assigned at birth.
* At least one of the following drawn within 30 days prior to pre-entry by any US laboratory that has a CLIA certification or its equivalent, or at any network-approved non-US laboratory that operates in accordance with Good Clinical Laboratory Practices (GCLP) and participates in appropriate external quality assurance programs:

  * Fasting plasma glucose 100-125 mg/dL (refer to the study protocol for a definition of fasting).
  * HbA1c between ≥5.7 and <6.5%
  * Homeostatic model assessment of insulin resistance (HOMA-IR) >3.0 (Refer to calculator: https://www.mdcalc.com/homa-ir-homeostatic-model-assessment-insulin-resistance)
* Documentation of negative hepatitis A virus (HAV) immunoglobulin M (IgM) or HAV vaccination prior to study entry.

  * NOTE: If documentation is not available prior to screening, this should be obtained through routine clinical care within 30 days prior to entry.
* Hepatic fat content (i.e., IHTG) ≥5%, as determined by liver magnetic resonance imaging-proton density fat fraction (MRI-PDFF) within 14 days prior to entry (and between 1-30 days after screening).

  * NOTE: Refer to the study protocol for more details.
* CD4+ T-cell count ≥200 cells/mm^3 within 30 days prior to pre-entry (may be from standard of care) at any US laboratory that has a CLIA certification or its equivalent, or at any network-approved non-US laboratory that is Immunology Quality Assurance (IQA) certified.
* The following laboratory values obtained within 30 days prior to pre-entry by any US laboratory that has a CLIA certification or its equivalent, or at any network-approved non-US laboratory that operates in accordance with GCLP and participates in appropriate external quality assurance programs:

  * Absolute neutrophil count (ANC) >750 cells/mm^3
  * Hemoglobin >10 g/dL for individuals assigned male at birth and >9 g/dL for individuals assigned female at birth
  * Creatinine clearance (CrCl) ≥50 mL/min, as calculated by the CKD-Epi equation.
  * NOTE: Please refer to A5371 protocol-specific web page (PSWP) for the website link to calculate CrCl using the CKD-Epi calculator.
  * NOTE: Calculations will be done without using cystatin C. Please refer to the A5371 Manual of Operating Procedures (MOPS) for further details.
  * Aspartate aminotransferase (AST) (SGOT) ≤3 x ULN on at least two measurements, with at least one within 30 days prior to pre-entry. Participants must also have no evidence of AST >3 x ULN within the 3 months prior to entry, from routine clinical monitoring, if available. If no additional monitoring is available in the 3 months prior to entry, additional testing should be obtained within the screening interval (2-4 weeks apart) to ensure stability.
  * Alanine aminotransferase (ALT) (SGPT) ≤3 x ULN on at least two measurements, with at least one within 30 days prior to pre-entry. Participants must also have no evidence of ALT >3 x ULN within the 3 months prior to entry, from routine clinical monitoring, if available. If no additional monitoring is available in the 3 months prior to entry, additional testing should be obtained within the screening interval (2-4 weeks apart) to ensure stability.
  * Fasting triglyceride level ≤500 mg/dL.
  * NOTE A: See the study protocol for a definition of fasting.
  * NOTE B: If level is >500 mg/dL, level may be rechecked within the screening window.
* For individuals taking daily medications with anti-inflammatory properties, including but not limited to, statins and chronic corticosteroids (inhaled corticosteroids exempt), the doses must be stable as determined by the site investigator for ≥3 months prior to study entry, and the individual should have no active plans to change dosing during the study period.
* For individuals taking daily lipid-lowering medications (such as statins, fibrates, niacin, fish oil), the doses must be stable as determined by the site investigator for ≥3 months prior to study entry, and the individual should have no active plans to change dosing during the study period.

  * NOTE: Lipid-lowering equivalents for niacin and fish oil are ≥1 g and ≥3 g daily, respectively.
* Ability and willingness of participant to provide informed consent
* Willingness and ability to use auto-inject pen weekly for 24 weeks.
* Willingness and ability to undergo MRI scans.

  * NOTE: Anxiolytics will not be provided through the study but may be provided at site expense.
* For persons able to become pregnant, a negative serum or urine pregnancy test (urine test must have a sensitivity of <25 mIU/mL) both 1) at screening (within 30 days prior to pre-entry MRI) and 2) within 3 days before or at entry (prior to registration into study) by any US clinic or laboratory that has a CLIA certification or its equivalent, or is using a point of care (POC)/ CLIA-waived test, or at any network-approved non-US laboratory or clinic that operates in accordance with Good Clinical Laboratory Practices (GCLP) and participates in appropriate external quality assurance programs.

  * NOTE: Individuals able to become pregnant are defined as individuals who have reached menarche and who have not been post-menopausal for at least 24 consecutive months (i.e., have had menses within the preceding 24 months), and have not undergone surgical sterilization such as hysterectomy, bilateral oophorectomy, tubal ligation, or salpingectomy.
* If participating in sexual activity that could lead to the participant becoming pregnant, the participant must agree to use contraception while on study drug (24 weeks) and for 2 months following the last dose of study drug. At least one of the following must be used:

  * Intrauterine device (IUD)
  * Hormone-based contraceptive
  * Partner sterilization (i.e., vasectomy) and is the sole partner for the participant.
  * NOTE: Participant self-report of partner sterilization is acceptable.
* For individuals taking Vitamin E (any dose), the dose must be stable as determined by the site investigator for more than 1 year prior to entry.
* Willingness to be contacted by telephone or e-mail by study staff throughout the study.

Exclusion Criteria:

* Known active hepatitis C virus (HCV) infection, defined as a detectable HCV RNA within 24 weeks prior to study entry.

  * NOTE A: Individuals with HCV RNA below the limit of quantitation for >24 weeks prior to study entry are eligible, i.e., individuals who have been treated for hepatitis C are eligible if they have completed therapy >24 weeks prior to study entry, and/or individuals who spontaneously cleared hepatitis C virus are eligible as long as they have had undetectable HCV RNA for >24 weeks. HCV RNA testing is not provided by the study.
  * NOTE B: If HCV antibody testing has not been performed in the 5 years prior to screening and the participant does not have history of cured HCV infection, HCV antibody testing should be repeated at screening. If screening HCV antibody is positive or reactive, the individual is not eligible and should be referred for clinical evaluation through routine care.
* Active/chronic hepatitis B (HBV), defined as a positive hepatitis B surface antigen (HBsAg) at screening.

  * NOTE A: HBsAg testing is only required at screening if HBV laboratory results are not available within the last 5 years prior to screening and individual does not have documented immunity.
  * NOTE B: If HBsAg positive, individual is not eligible and should be referred for clinical evaluation through routine care.
* Known active severe delayed gastric emptying, as determined by the site investigator.
* Gain or loss of >5% body weight within 12 weeks prior to study entry.

  * NOTE: Self-report recall is acceptable.
* Any plans to change diet or exercise regimen significantly, except for the adoption of study provided suggestions for diet and exercise, within the study period.

  * NOTE: "Significantly" refers to intent to join a weight-loss program such as Weight Watchers, or start a specific diet (such as ketogenic or very low carbohydrate).
* Known acute or chronic liver disease with cirrhosis or portal hypertension.
* History of liver transplant.
* Breastfeeding or plans to become pregnant.
* Current diagnosis of diabetes mellitus or current use of diabetes medications, or a laboratory measurement of hemoglobin A1c ≥6.5% at screening.

  * NOTE: Stable use of metformin (i.e., for ≥12 weeks) for indication other than diabetes (e.g., polycystic ovarian syndrome or pre-diabetes/impaired fasting glucose) may be permitted with approval of the Clinical Management Committee (CMC).
* Known retinopathy (excluding remote history of cotton wool spots).
* Personal or family (first-degree relative) history of medullary thyroid carcinoma or multiple endocrine neoplasia type 2 (MEN2).
* Untreated, poorly controlled, or previously undiagnosed thyroid disease defined as the presence of abnormal thyroid-stimulating hormone (TSH) at screening with no clear explanation.
* Unexplained hypercalcemia corrected for albumin that is >10.5 mg/dL at screening. Please refer to the A5371 MOPS for the calculation.
* Use of any immunomodulatory (including prednisone equivalent of ≥10 mg), HIV vaccine, investigational therapy, or TNF-α therapy within 3 months prior to study entry.
* Use of human growth hormone, tesamorelin, supraphysiologic testosterone to achieve therapeutic blood levels, or any use of other anabolic steroids within 3 months prior to study entry or plans to start these while on study.

  * NOTE: Chronic, stable hormone replacement therapy ≥3 months prior to entry in men with diagnosed hypogonadism or transgender person on masculinizing hormonal therapy is permitted.
* Use of estrogens or progesterones at supraphysiologic doses within 3 months prior to study entry.

  * NOTE: Stable doses used for contraception, post-menopausal hormone replacement or feminizing hormone therapy for transgender persons ≥3 months prior to entry is permitted.
* Known allergy/sensitivity or any hypersensitivity to components of study drug or its formulation.
* Current serious illness requiring systemic treatment and/or hospitalization.

  * NOTE: The individual can be rescreened when they complete therapy or are clinically stable as determined by the site investigator.
* Use of GLP-1 agonists within 24 weeks prior to study entry.
* Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
* Excessive consumption of alcohol of ≥3 months within 90 days prior to screening, defined as:

  * Consuming ≥5 alcoholic drinks for men or consuming ≥4 alcoholic drinks for women during a single occasion (i.e., at the same time or within a couple of hours of each other), or
  * ≥3 drinks on 4 or more days of the week on average for men or ≥2 drinks on 4 or more days of the week on average for women.
  * NOTE: For transgender study participants, sites should use the parameter that matches sex assigned at birth.
* Known chronic pancreatitis or more than one episode of pancreatitis ever in the past.
* Inability to keep study product at 36°F to 46°F (2°C to 8°C) prior to first use, or to maintain the study product at a controlled room temperature between 59°F and 86°F (15°C to 30°C) following first use.
* Intent to use any medication likely to cause significant changes in weight during the study period.

  * NOTE: Refer to the study protocol for a list of medications in this category.
* Use of stavudine within 12 months prior to study entry.
* Prior bariatric surgery (e.g., lap band, gastric sleeve, or Roux-en-Y bypass surgery) or major gastric surgery or plans to undergo weight reduction surgery while on study.
* Individuals with any metal, implantable devices (e.g., pacemakers, prosthetics), or shrapnel, per standard MRI exclusion criteria.
* Any condition that the site investigator believes would make the individual unsuitable for participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2021-02-19 (Actual); Primary Completion 2023-03-16 (Actual); Study Completion 2023-09-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristine Erlandson, MD, MS, Study Chair — University of Colorado Hospital CRS; Jordan E. Lake, MD, MSc, Study Chair — Houston AIDS Research Team CRS
Locations (9):
- United States (8):
  - Alabama CRS (Site ID: 31788), Birmingham, Alabama
  - University of Colorado Hospital CRS (Site ID: 6101), Aurora, Colorado
  - Johns Hopkins University CRS, Baltimore, Maryland
  - Massachusetts General Hospital CRS (MGH CRS) (Site ID: 101), Boston, Massachusetts
  - Cincinnati Clinical Research Site (Site ID: 2401), Cincinnati, Ohio
  - Ohio State University CRS (Site ID: 2301), Columbus, Ohio
  - Houston AIDS Research Team CRS (Site ID: 31473), Houston, Texas
  - University of Washington AIDS CRS (Site ID: 1401), Seattle, Washington
- Instituto de Pesquisa Clinica Evandro Chagas (IPEC) CRS (Site ID: 12101), Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie results in the publication, after deidentification.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months following publication and available throughout period of funding of the AIDS Clinical Trials Group by NIH.
Access Criteria: * With whom?
    * Researchers who provide a methodologically sound proposal for use of the data that is approved by the AIDS Clinical Trials Group.
  * For what types of analyses?
    * To achieve aims in the proposal approved by the AIDS Clinical Trials Group.
  * By what mechanism will data be made available?
    * Researchers may submit a request for access to data using the AIDS Clinical Trials Group "Data Request" form at: https://submit.mis.s-3.net/ Researchers of approved proposals will need to sign an AIDS Clinical Trials Group Data Use Agreement before receiving the data.

REFERENCES:
- [Derived] Corley M, Pang A, Kitch D, Kantor A, Sattler F, Belaunzaran-Zamudio P, Brown T, Landay A, Lake J, Erlandson K. Epigenetic Aging and Treatment Response to Semaglutide in the SLIM LIVER Study. Res Sq [Preprint]. 2025 Oct 1:rs.3.rs-7697256. doi: 10.21203/rs.3.rs-7697256/v1. PMID 41256006
- [Derived] Ditzenberger GL, Lake JE, Kitch DW, Kantor A, Muthupillai R, Moser C, Belaunzaran-Zamudio PF, Brown TT, Corey K, Landay AL, Avihingsanon A, Sattler FR, Erlandson KM. Effects of Semaglutide on Muscle Structure and Function in the SLIM LIVER Study. Clin Infect Dis. 2025 Feb 24;80(2):389-396. doi: 10.1093/cid/ciae384. PMID 39046173
- See also: The Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), corrected Version 2.1, July 2017. — https://rsc.niaid.nih.gov/clinical-research-sites/daids-adverse-event-grading-tables
- See also: Manual for Expedited Reporting of Adverse Events to DAIDS (DAIDS EAE Manual), Version 2.0, January 2010. — http://rsc.niaid.nih.gov/clinical-research-sites/manual-expedited-reporting-adverse-events-daids

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first participant was enrolled in February 2021. Study enrollment was completed in September 2022 with the enrollment of the last participant. Participants were enrolled from 9 sites in the United States and Brazil.
Period: Overall Study
Arm/Group | Semaglutide
Started | 51
Completed Study Treatment | 48
Completed | 47
Not Completed | 4
Not completed — Withdrawal by Subject | 2
Not completed — Protocol Violation | 1
Not completed — Incarceration | 1

BASELINE CHARACTERISTICS:
Population: All participants who were enrolled to the study.
Arm/Group | Semaglutide
Number analyzed (Participants) | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 48
  >=65 years | 3
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 52 [41 to 58]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Cisgender Male | 30
  Cisgender Female | 18
  Transgender Female | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20
  Not Hispanic or Latino | 31
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 16
  White | 30
  More than one race | 1
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 49
  Brazil | 2
Intra-Hepatic Triglyceride Content (IHTG) [Mean (Standard Deviation); unit: percent of IHTG content] — IHTG (a type of fat stored in the liver) was quantified by magnetic resonance imaging-proton density fat fraction (MRI-PDFF). Population: All participants who remained on study treatment until 28 days prior to the Week 24 MRI and who did not start prohibited medications known to cause changes in weight prior to the Week 24 MRI.
  percent of IHTG content
    number analyzed (Participants) | 48
    (all) | 12.7 (6.05)

OUTCOME MEASURES:

1. Primary Outcome: Change (Absolute) in IHTG (%)
Description: The absolute change in intra-hepatic triglyceride content (%), as quantfied by MRI-PDFF, from the pre-entry visit to the Week 24 visit.
Time Frame: Measured at pre-entry and Week 24
Population: Analysis was done in the per-protocol population. These were all participants who remained on study treatment until 28 days prior to the Week 24 MRI and who did not start prohibited medications known to cause changes in weight prior to the Week 24 MRI.
Measure: Mean (95% Confidence Interval); unit: IHTG %
Arm/Group | Semaglutide
Number analyzed (Participants) | 48
IHTG % | -4.24 [-5.41 to -3.06]
Statistical Analysis 1: Comparison: Semaglutide; The study was powered to detect an absolute IHTG change of -5% assuming a null change of 0%, a standard deviation of absolute IHTG change of 9%, and 37 evaluable participants; Test type: Other — This was a single arm trial; p < 0.001, Regression, Linear; Mean Difference (Net) = -4.24, 95% CI 2-sided [-5.41 to -3.06], Standard Deviation 4.05

2. Secondary Outcome: Change (Percent) in IHTG (%)
Description: The percentage change in intra-hepatic triglyceride content (%), as quantfied by MRI-PDFF, from the pre-entry visit to the Week 24 visit. The percentage change is defined as IHTC % at week 24 minus IHTC % at pre-entry, then divided by IHTC % at pre-entry, then multiplied by 100.
Time Frame: Measured at pre-entry and Week 24
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Relative change %
Arm/Group | Semaglutide
Number analyzed (Participants) | 48
Relative change % | -31.33 [-39.04 to -23.62]
Statistical Analysis 1: Comparison: Semaglutide; Test type: Other — This was a single arm trial; p < 0.001, Regression, Linear — No adjustment for multiple comparisons; Mean Difference (Net) = -31.33, 95% CI 2-sided [-39.04 to -23.62], Standard Deviation 26.5

3. Secondary Outcome: Level of IHTG (%)
Description: Intra-hepatic triglyceride content (%) at Week 24 (<5% vs. >=5%). All participants were >=5% at pre-entry.
Time Frame: Measured at Week 24
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Semaglutide
Number analyzed (Participants) | 48
participants
  <5% IHTG | 14
  >=5% IHTG | 34

4. Secondary Outcome: Occurrence of Premature Discontinuation of Study Treatment
Description: Premature study treatment discontinuation prior to the Week 24 visit.
Time Frame: Measured through Week 24
Population: Analysis was done in the intent-to-treat population. These were all participants who were enrolled to the study.
Measure: Number; unit: participants
Arm/Group | Semaglutide
Number analyzed (Participants) | 51
participants
  Premature discontinuation | 3
  Completed study treatment | 48

5. Secondary Outcome: Occurrence of Grade ≥3 Adverse Event That is Related to Study Treatment
Description: Graded according to the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), corrected Version 2.1, July 2017. Adverse events are graded on a scale from 1-5: 1=mild, 2=moderate, 3=severe, 4=life-threatening, 5=death.
Time Frame: Measured through Week 24
Population: Analysis was done in the intent-to-treat population. These were all participants who were enrolled to the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide
Number analyzed (Participants) | 51
Participants
  Yes | 2
  No | 49

6. Secondary Outcome: Change (Absolute) in Body Mass Index (BMI)
Description: The absolute change in body mass index from the study entry (Week 0) visit to the Week 24 visit.
Time Frame: Measured at Week 0 and Week 24
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: kg/m^2
Arm/Group | Semaglutide
Number analyzed (Participants) | 49
kg/m^2 | -2.77 [-3.36 to -2.17]
Statistical Analysis 1: Comparison: Semaglutide; Test type: Other — This was a single arm trial; p < 0.001, Regression, Linear — Not adjusted for multiple comparisons; Mean Difference (Net) = -2.77, 95% CI 2-sided [-3.36 to -2.17], Standard Deviation 2.05

7. Secondary Outcome: Change (Absolute) in Body Mass Index (BMI)
Description: The absolute change in body mass index from the study entry (Week 0) visit to the Week 12 visit.
Time Frame: Measured from Week 0 to Week 12
Population: Per-protocol population (N=49)
Measure: Mean (95% Confidence Interval); unit: kg/m^2
Arm/Group | Semaglutide
Number analyzed (Participants) | 49
kg/m^2 | -2.15 [-2.55 to -1.75]
Statistical Analysis 1: Comparison: Semaglutide; Test type: Other — This was a single arm trial; p < 0.001, Regression, Linear — Not adjusted for multiple comparisons; Mean Difference (Net) = -2.15, 95% CI 2-sided [-2.55 to -1.75], Standard Deviation 1.38

8. Secondary Outcome: Change (Absolute) in Body Weight
Description: The absolute change in body weight from the study entry (Week 0) visit to the Week 24 visit.
Time Frame: Measured at Week 0 and Week 24
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: kg
Arm/Group | Semaglutide
Number analyzed (Participants) | 48
kg | -7.80 [-9.48 to -6.13]
Statistical Analysis 1: Comparison: Semaglutide; Test type: Other — This was a single arm trial; p < 0.001, Regression, Linear — Not adjusted for multiple comparisons; Mean Difference (Net) = -7.80, 95% CI 2-sided [-9.48 to -6.13], Standard Deviation 5.77

9. Secondary Outcome: Change (Absolute) in Body Weight
Description: The absolute change in body weight from the study entry (Week 0) visit to the Week 12 visit.
Time Frame: Measured at Week 0 and Week 12
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: kg
Arm/Group | Semaglutide
Number analyzed (Participants) | 49
kg | -6.16 [-7.30 to -5.03]
Statistical Analysis 1: Comparison: Semaglutide; Test type: Other — This was a single arm trial; p < 0.001, Regression, Linear — Not adjusted for multiple comparisons; Mean Difference (Net) = -6.16, 95% CI 2-sided [-7.30 to -5.03], Standard Deviation 3.96

10. Secondary Outcome: Change (Absolute) in Minimum Waist Circumference (WC)
Description: The absolute change in minimum WC from the study entry (Week 0) visit to the Week 24 visit.
Time Frame: Measured at Week 0 and Week 24
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: cm
Arm/Group | Semaglutide
Number analyzed (Participants) | 48
cm | -6.66 [-8.54 to -4.78]
Statistical Analysis 1: Comparison: Semaglutide; Test type: Other — This was a single arm trial; p < 0.001, Regression, Linear — Not adjusted for multiple comparisons; Mean Difference (Net) = -6.66, 95% CI 2-sided [-8.54 to -4.78], Standard Deviation 6.47

11. Secondary Outcome: Change (Absolute) in Minimum Waist Circumference (WC)
Description: The absolute change in minimum WC from the study entry (Week 0) visit to the Week 12 visit.
Time Frame: Measured at Week 0 and Week 12
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: cm
Arm/Group | Semaglutide
Number analyzed (Participants) | 48
cm | -5.53 [-7.07 to -3.99]
Statistical Analysis 1: Comparison: Semaglutide; Test type: Other — This was a single arm trial; p < 0.001, Regression, Linear — Not adjusted for multiple comparisons; Mean Difference (Net) = -5.53, 95% CI 2-sided [-7.07 to -3.99], Standard Deviation 5.30

12. Secondary Outcome: Change (Absolute) in Insulin Resistance (HOMA-IR)
Description: The absolute change in HOMA-IR from the study entry (Week 0) visit to the Week 24 visit.
  HOMA-IR (Homeostatic Model Assessment of Insulin Resistance) is a method used to estimate how well your body responds to insulin.
  HOMA-IR is caluclated with the following formula:
  (fasting glucose in mmol/L x fasting insulin in mIU/mL)/22.5
  A higher HOMA-IR score indicates a greater likelihood of insulin resistance.
Time Frame: Measured at Week 0 and Week 24
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: uU/ml*mmol/l/22.5
Arm/Group | Semaglutide
Number analyzed (Participants) | 47
uU/ml*mmol/l/22.5 | -1.46 [-3.17 to 0.25]
Statistical Analysis 1: Comparison: Semaglutide; Test type: Other — This was a single arm trial; p = 0.092, Regression, Linear — Not adjusted for multiple comparisons; Mean Difference (Net) = -1.46, 95% CI 2-sided [-3.17 to 0.25], Standard Deviation 5.82

13. Secondary Outcome: Change (Absolute) in Insulin Resistance (HOMA-IR)
Description: The absolute change in HOMA-IR from the study entry (Week 0) visit to the Week 12 visit.
  HOMA-IR (Homeostatic Model Assessment of Insulin Resistanc) is a method used to estimate how well your body responds to insulin.
  HOMA-IR is caluclated with the following formula:
  (fasting glucose in mmol/L x fasting insulin in mIU/mL)/22.5 A higher HOMA-IR score indicates a greater likelihood of insulin resistance.
Time Frame: Measured at Week 0 and Week 12
Population: Outcomes not available because fasting insulin data was not collected at Week 12.
Arm/Group | Semaglutide
Number analyzed (Participants) | 0

14. Secondary Outcome: Change (Absolute) in Hemoglobin A1C (HbA1c)
Description: The absolute change in HbA1c from the study entry (Week 0) visit to the Week 24 visit.
Time Frame: Measured at Week 0 and Week 24
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: HbA1c %
Arm/Group | Semaglutide
Number analyzed (Participants) | 48
HbA1c % | -0.25 [-0.32 to -0.17]
Statistical Analysis 1: Comparison: Semaglutide; Test type: Other — This was a single arm trial; p < 0.001, Regression, Linear — Not adjusted for multiple comparisons; Mean Difference (Net) = -0.25, 95% CI 2-sided [-0.32 to -0.17], Standard Deviation 0.259

15. Secondary Outcome: Change (Absolute) in Fasting Glucose
Description: The absolute change in fasting glucose from the study entry (Week 0) visit to the Week 24 visit.
Time Frame: Measured at Week 0 and Week 24
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: mg/dl
Arm/Group | Semaglutide
Number analyzed (Participants) | 48
mg/dl | -9.90 [-14.70 to -5.09]
Statistical Analysis 1: Comparison: Semaglutide; Test type: Other — This was a single arm trial; p < 0.001, Regression, Linear — Not adjusted for multiple comparisons; Mean Difference (Net) = -9.90, 95% CI 2-sided [-14.70 to -5.09], Standard Deviation 16.6

16. Secondary Outcome: Change (Absolute) in Fasting Glucose
Description: The absolute change in fasting glucose from the study entry (Week 0) visit to the Week 12 visit.
Time Frame: Measured at Week 0 and Week 12
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: mg/dl
Arm/Group | Semaglutide
Number analyzed (Participants) | 47
mg/dl | -8.87 [-12.26 to -5.48]
Statistical Analysis 1: Comparison: Semaglutide; Test type: Other — This was a single arm trial; p < 0.001, Regression, Linear — Not adjusted for multiple comparisons; Mean Difference (Net) = -8.87, 95% CI 2-sided [-12.26 to -5.48], Standard Deviation 11.5

17. Secondary Outcome: Change (Absolute) in Fasting Total Cholesterol
Description: The absolute change in fasting total cholesterol from the study entry (Week 0) visit to the Week 24 visit.
Time Frame: Measured at Week 0 and Week 24
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: mg/dl
Arm/Group | Semaglutide
Number analyzed (Participants) | 46
mg/dl | -3.98 [-10.84 to 2.89]
Statistical Analysis 1: Comparison: Semaglutide; Test type: Other — This was a single arm trial; p = 0.25, Regression, Linear — Not adjusted for multiple comparisons; Mean Difference (Net) = -3.98, 95% CI 2-sided [-10.84 to 2.89], Standard Deviation 23.1

18. Secondary Outcome: Change (Absolute) in Fasting Total Cholesterol
Description: The absolute change in fasting total cholesterol from the study entry (Week 0) visit to the Week 12 visit.
Time Frame: Measured at Week 0 and Week 12
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: mg/dl
Arm/Group | Semaglutide
Number analyzed (Participants) | 46
mg/dl | -11.93 [-19.79 to -4.08]
Statistical Analysis 1: Comparison: Semaglutide; Test type: Other — This was a single arm trial; p = 0.004, Regression, Linear — Not adjusted for multiple comparisons; Mean Difference (Net) = -11.93, 95% CI 2-sided [-19.79 to -4.08], Standard Deviation 26.4

19. Secondary Outcome: Change (Absolute) in Fasting LDL Cholesterol
Description: The absolute change in fasting LDL cholesterol from the study entry (Week 0) visit to the Week 24 visit.
Time Frame: Measured at Week 0 and Week 24
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: mg/dl
Arm/Group | Semaglutide
Number analyzed (Participants) | 46
mg/dl | -1.04 [-7.14 to 5.05]
Statistical Analysis 1: Comparison: Semaglutide; Test type: Other — This was a single arm trial; p = 0.73, Regression, Linear — Not adjusted for multiple comparisons; Mean Difference (Net) = -1.04, 95% CI 2-sided [-7.14 to 5.05], Standard Deviation 20.5

20. Secondary Outcome: Change (Absolute) in Fasting LDL Cholesterol
Description: The absolute change in fasting LDL cholesterol from the study entry (Week 0) visit to the Week 12 visit.
Time Frame: Measured at Week 0 and Week 12
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: mg/dl
Arm/Group | Semaglutide
Number analyzed (Participants) | 45
mg/dl | -6.91 [-13.85 to 0.03]
Statistical Analysis 1: Comparison: Semaglutide; Test type: Other — This was a single arm trial; p = 0.051, Regression, Linear — Not adjusted for multiple comparisons; Mean Difference (Net) = -6.91, 95% CI 2-sided [-13.85 to 0.03], Standard Deviation 23.1

21. Secondary Outcome: Change (Absolute) in Fasting HDL Cholesterol
Description: The absolute change in fasting HDL cholesterol from the study entry (Week 0) visit to the Week 24 visit.
Time Frame: Measured at Week 0 and Week 24
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: mg/dl
Arm/Group | Semaglutide
Number analyzed (Participants) | 46
mg/dl | 2.04 [-0.02 to 4.11]
Statistical Analysis 1: Comparison: Semaglutide; Test type: Other — This was a single arm trial; p = 0.053, Regression, Linear — Not adjusted for multiple comparisons; Mean Difference (Net) = 2.04, 95% CI 2-sided [-0.02 to 4.11], Standard Deviation 6.96

22. Secondary Outcome: Change (Absolute) in Fasting HDL Cholesterol
Description: The absolute change in fasting HDL cholesterol from the study entry (Week 0) visit to the Week 12 visit.
Time Frame: Measured at Week 0 and Week 12
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: mg/dl
Arm/Group | Semaglutide
Number analyzed (Participants) | 46
mg/dl | -0.78 [-2.76 to 1.20]
Statistical Analysis 1: Comparison: Semaglutide; Test type: Other — This was a single arm trial; p = 0.43, Regression, Linear — Not adjusted for multiple comparisons; Mean Difference (Net) = -0.78, 95% CI 2-sided [-2.76 to 1.20], Standard Deviation 6.66

23. Secondary Outcome: Change (Absolute) in Fasting Triglycerides
Description: The absolute change in fasting triglycerides from the study entry (Week 0) visit to the Week 24 visit.
Time Frame: Measured at Week 0 and Week 24
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: mg/dl
Arm/Group | Semaglutide
Number analyzed (Participants) | 46
mg/dl | -26.78 [-46.04 to -7.53]
Statistical Analysis 1: Comparison: Semaglutide; Test type: Other — This was a single arm trial; p = 0.007, Regression, Linear — Not adjusted for multiple comparisons; Mean Difference (Net) = -26.78, 95% CI 2-sided [-46.04 to -7.53], Standard Deviation 64.8

24. Secondary Outcome: Change (Absolute) in Fasting Triglycerides
Description: The absolute change in fasting triglycerides from the study entry (Week 0) visit to the Week 12 visit.
Time Frame: Measured at Week 0 and Week 12
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: mg/dl
Arm/Group | Semaglutide
Number analyzed (Participants) | 46
mg/dl | -18.65 [-33.29 to -4.01]
Statistical Analysis 1: Comparison: Semaglutide; Test type: Other — This was a single arm trial; p = 0.014, Regression, Linear — Not adjusted for multiple comparisons; Mean Difference (Net) = -18.65, 95% CI 2-sided [-33.29 to -4.01], Standard Deviation 49.3

25. Secondary Outcome: Presence of Metabolic Syndrome
Description: Metabolic syndrome is defined as having ≥3 of the following: increased minimum WC (>=40 inches for male sex at birth; >=35 inches for female sex at birth), increased fasting triglyceride level (>150 mg/dL or taking lipid-lowering medication), reduced fasting HDL cholesterol (<40 mg/dL for male sex at birth; <50 mg/dL for female sex at birth), increased blood pressure (>=135/85 mmHg or taking BP medication), and increased fasting glucose (>100 mg/dL or taking glucose-lowering medication).
Time Frame: Measured at Weeks 0, 12 and 24
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide
Number analyzed (Participants) | 49
Participants
  Baseline: Metabolic syndrome | 38
  Baseline: No metabolic syndrome | 11
  Week 12: number analyzed (Participants) | 46
  Week 12: Metabolic syndrome | 25
  Week 12: No metabolic syndrome | 21
  Week 24: number analyzed (Participants) | 47
  Week 24: Metabolic syndrome | 28
  Week 24: No metabolic syndrome | 19
Statistical Analysis 1: Comparison: Semaglutide; Comparison between Baseline and Week 12; Test type: Other — This was a single arm trial; p = 0.016, GEE model for repeated binary outcomes — Not adjusted for multiple comparisons; The GEE model used a log link and an unstructured correlation; Risk Ratio (RR) = 0.72, 95% CI 2-sided [0.55 to 0.94] — The risk ratio is comparing the estimated risk at Week 12 (0.55; 95% CI: 0.43, 0.72) to estimated risk at Baseline (0.77; 95% CI: 0.67, 0.90)
Statistical Analysis 2: Comparison: Semaglutide; Comparison between Baseline and Week 24; Test type: Other — This was a single arm trial; p = 0.033, GEE model for repeated binary outcomes — Not adjusted for multiple comparisons; The GEE model used a log link and an unstructured correlation; Risk Ratio (RR) = 0.75, 95% CI 2-sided [0.58 to 0.98] — The risk ratio is comparing the estimated risk at Week 24 (0.58; 95% CI: 0.46, 0.74) to estimated risk at Baseline (0.77; 95% CI: 0.67, 0.90)

ADVERSE EVENTS:
Time Frame: From study entry to study completion at Week 48 or premature study discontinuation.
Description: All AEs must be recorded on the eCRFs if any of the following criteria have been met:
  * All Grade ≥3 AEs
  * Grade ≥2 laboratory values
  * All AEs that led to a change in study treatment/intervention regardless of grade
  * All AEs meeting SAE definition or EAE reporting requirement
Groups:
- Semaglutide: All participants will receive a dose of 0.25 mg of semaglutide weekly starting at study entry, followed by 0.5 mg weekly starting at Week 2, and then 1.0 mg weekly from Weeks 4 through 24.
  Semaglutide: Administered subcutaneously
Arm/Group | Semaglutide
All-Cause Mortality (participants affected / at risk) | 0/51
Serious Adverse Events (participants affected / at risk) | 2/51
Other Adverse Events (participants affected / at risk) | 20/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Semaglutide (N=51)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Serotonin syndrome (Nervous system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Semaglutide (N=51)
Abdominal pain (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 2
Chills (General disorders) | 1
Fatigue (General disorders) | 1
Blood cholesterol increased (Investigations) | 1
Blood creatinine increased (Investigations) | 2
Blood glucose increased (Investigations) | 2
Blood phosphorus decreased (Investigations) | 1
Blood triglycerides increased (Investigations) | 2
Blood uric acid increased (Investigations) | 1
Creatinine renal clearance decreased (Investigations) | 6
Creatinine renal clearance increased (Investigations) | 1
Haemoglobin decreased (Investigations) | 1
Lipids increased (Investigations) | 1
Platelet count decreased (Investigations) | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1
Serotonin syndrome (Nervous system disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-06-22): https://cdn.clinicaltrials.gov/large-docs/89/NCT04216589/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-23): https://cdn.clinicaltrials.gov/large-docs/89/NCT04216589/SAP_001.pdf